CLINICAL TRIAL: NCT01657669
Title: Short-term Clinical Effects of Intravitreal Aflibercept Injection 2.0mg as a Predictor of Long-term Results
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Retina Research Institute, LLC (Other)
Collaborators: Valley Retina Institute (Other)
Responsible Party: Principal Investigator, Rhonda Weeks, Gaurav K. Shah, MD, Principal Investigator, Retina Research Institute, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-01-12
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Age Related Macular Degeneration
Keywords: Choroidal neovascularization due to AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravitreal Aflibercept injection (Other): Intravitreal Aflibercept injection 2.0 mg dosed every 4 weeks (monthly) for the first 3 months followed by 2.0 mg (0.05mg) via intravitreal injection once every 8 weeks (2 months).
  Interventions: Drug: Intravitreal Aflibercept injection

INTERVENTIONS:
Drug: Intravitreal Aflibercept injection — Intravitreal Aflibercept injection 2.0 mg dosed every 4 weeks (monthly) for the first 3 months followed by 2.0 mg (0.05mL) via intravitreal injection once every 8 weeks (2 months). Dosing at monthly intervals is allowed if needed in the opinion of the investigator based on presence of fluid on OCT and/or a decrease in visual acuity of 5 letters or more from the best previous visit.

SUMMARY:
This is an open label study to evaluate 2.0 mg intravitreal aflibercept injection administered in subject who have active choroidal neovascularization due to Age Related Macular Degeneration (AMD).

DETAILED DESCRIPTION:
Twenty (20) consented participant who meet the inclusion criteria will be enrolled to be followed for 48 weeks. All subjects will receive 2.0 mg intravitreal aflibercept injections with three initial monthly doses, and mandatory doses at Weeks 16, 24, 32, and 40. Dosing at monthly intervals is allowed if needed in the opinion of the investigator based on presence of fluid on Optical Coherence Tomography (OCT) and/or a decrease in visual acuity of greater than or equal to 5 letters from the best previous visit. Only one eye will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

Ability to provide written informed consent and comply with study assessments for the full duration of the study.

Age 50 years and above.

Choroidal neovascularization secondary to AMD with central retinal thickness greater than or equal to 300um.

Best corrected visual acuity in the study eye between 20/40 and 20/400 using an ETDRS chart -

Exclusion Criteria:

Pregnancy (positive urine pregnancy test) or lactation.

Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.

Participation in a study or an investigational drug or device within the past 30 days prior to enrolling in the study.

Presence of significant subfoveal fibrosis or atrophy.

Previously treated subjects:

Prior treatment with anti-VEGF therapy in the study eye within 28 days of baseline More than six (6) prior treatments with anti-VEGF therapy in the study eye within 1 year.

Prior treatment with PDT within the past 3 months or more than 2 prior PDT treatments.

Prior treatment with intravitreal aflibercept injection Prior treatment with triamcinolone in the study eye within 6 months of baseline.

Prior treatment with dexamethasone in the study eye within 30 days prior to baseline.

Intraocular surgery (including cataract surgery)in the study eye within 2 months preceding baseline

History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in the study eye.

Active intraocular inflammation (grade trace or above) in the study eye

Current vitreous hemorrhage in the study eye

History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye.

Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye.

Uncontrolled glaucoma in the study eye (defined as IOP greater than or equal to 30 mmHg despite treatment with anti-glaucoma medication)

History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 3 months of study enrollment.

History of allergy to fluorescein, ICG or iodine, not amenable to treatment

History of retinal pigment epithelial tear or rip.

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Resolution time of intraretinal cysts and sub retinal fluid on OCT | 12 months

SECONDARY OUTCOMES:
Mean change in OCT central foveal thickness | 12 months
The percentage of subjects with no fluid on OCT | 12 months
The percentage of subjects who lose less than 15 letters of visual acuity | 12 months
The percentage of subjects who gain greater than or equal to 15 letters of visual acuity | 12 months
Mean change in visual acuity | 12 months
Mean change in macular volume | 12 months
Quantitative change in area (microns) from baseline in choroidal neovascular lesion characteristics/size as measured by ICG/FA/Fundus photos | 12 months
Mean number of injections of 2.0 mg intravitreal aflibercept injection | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav K. Shah, MD, Principal Investigator — The Retina Institute
Locations (2):
- United States (2):
  - The Retina Institute, St Louis, Missouri
  - Valley Retina Institute, McAllen, Texas

REFERENCES:
- [Derived] Liu EM, Shah G, Blinder KJ, Smith BT, Thomas MA. Intravitreal Aflibercept for Neovascular AMD: Short-Term Clinical Effects of Intravitreal Aflibercept Injection as a Predictor of Long-Term Results. Ophthalmic Surg Lasers Imaging Retina. 2015 Nov-Dec;46(10):1021-7. doi: 10.3928/23258160-20151027-06. PMID 26599244